CLINICAL TRIAL: NCT04556513
Title: Functional Recovery From Acute Respiratory Distress Syndrome (ARDS) Due to COVID-19: Influence of Socio-Economic Status
Acronym: RECOVIDS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: QUENOT 2020
Record Dates: First submitted 2020-09-16; First posted 2020-09-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Covid19; ARDS; Functional Recovery
MeSH Terms: conditions — COVID-19 | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient: Patient hospitalized in ICU for PCR-proven SARS-COV-2 infection
  Interventions: Other: Paraclinical examination; Other: Clinical Examination; Other: Semi-directive interview; Other: quality of life questionnaires

INTERVENTIONS:
Other: Paraclinical examination — Respiratory functional tests
Other: Clinical Examination — Clinical Examination
Other: Semi-directive interview — By phone
Other: quality of life questionnaires — SF36, VSRQ, IESR, HADS

SUMMARY:
In this study, the investigators are attempting to evaluate the influence of socio-economic factors on the functional recovery (physical and psychological) of patients who developed ARDS after a COVID-19 infection, with the aim of offering personalized medical and social follow-up and support measures in order to avoid medium- and long-term complications, which can result in handicaps, reduced quality of life, and a higher risk of death.

ELIGIBILITY:
Inclusion Criteria:

* Inpatient in ICU for PCR-proven SARS-VOC-2 infection regardless of specimen type
* Patient who received a chest CT scan in the initial phase of management (either just before or during hospitalization in the intensive care unit)
* Patient who has received invasive or non-invasive ventilatory support, or humidified and heated high-flow oxygen (HFO).
* ARDS meeting the criteria of the 2012 Berlin definition. For patients who have received only HFO, a flow rate at least equal to 50L/minute with a FiO2 strictly greater than 50% with a PaO2/FiO2 ratio less than or equal to 200 will be required for inclusion.
* Patient who gave oral consent after being informed about the conduct of this study.

Exclusion Criteria:

* Patient with limited autonomy prior to hospitalization in limited intensive care unit: walking distance of less than 50 meters, WHO classification status 3 and 4.
* Patient with a history of chronic respiratory failure as defined by the use of long-term oxygen therapy or non-invasive home ventilation, excluding patients with SAS and/or hypoventilation obesity syndrome.
* Patient with a history of central or peripheral neurological conditions limiting the patient's motor autonomy and the performance on gait tests or Pulmonary function Tests
* Patient refusing to participate
* Patient < 18 years of age
* Patient not affiliated or not benefiting from national health insurance
* Patient under guardianship, curatorship or protected adult
* Patient unable to understand and consent to the research protocol

SECONDARY EXCLUSION CRITERIA

* Patient not showing up for visit at M6
* Patients who have not had all the examinations necessary to evaluate the main endpoint (Spirometry, DLCO, TM6 and CT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who has been managed in intensive care for covid-19 infection.
Sampling Method: Non-Probability Sample
Enrollment: 543 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Respiratory sequelae 6 months after resuscitation. | Through study completion, an average of 6 months
  Defined by the presence of at least one of the following :
  * An alteration of the alveolar-capillary diffusion of CO <80% of the predicted normal values
  * And/or a forced vital capacity <80% of predicted normal values
  * and/or O2 desaturation in the 6-minute walk test
  * And/or pulmonary parenchymatous disease with fibrosis in tomodensitometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Declercq PL, Fournel I, Demeyere M, Berraies A, Ksiazek E, Nyunga M, Daubin C, Ampere A, Sauneuf B, Badie J, Delbove A, Nseir S, Artaud-Macari E, Bironneau V, Ramakers M, Maizel J, Miailhe AF, Lacombe B, Delberghe N, Oulehri W, Georges H, Tchenio X, Clarot C, Redureau E, Bourdin G, Federici L, Adda M, Schnell D, Bousta M, Salmon-Gandonniere C, Vanderlinden T, Plantefeve G, Delacour D, Delpierre C, Le Bouar G, Sedillot N, Beduneau G, Riviere A, Meunier-Beillard N, Gelinotte S, Rigaud JP, Labruyere M, Georges M, Binquet C, Quenot JP; RECOVIDS trial investigators, the CRICS-TRIGGERSEP, BOREAL research networks. Influence of socio-economic status on functional recovery after ARDS caused by SARS-CoV-2: the multicentre, observational RECOVIDS study. Intensive Care Med. 2023 Oct;49(10):1168-1180. doi: 10.1007/s00134-023-07180-y. Epub 2023 Aug 24. PMID 37620561
- [Derived] Declercq PL, Fournel I, Demeyere M, Ksiazek E, Meunier-Beillard N, Riviere A, Clarot C, Maizel J, Schnell D, Plantefeve G, Ampere A, Daubin C, Sauneuf B, Kalfon P, Federici L, Redureau E, Bousta M, Lagache L, Vanderlinden T, Nseir S, La Combe B, Bourdin G, Monchi M, Nyunga M, Ramakers M, Oulehri W, Georges H, Salmon Gandonniere C, Badie J, Delbove A, Monnet X, Beduneau G, Artaud-Macari E, Abraham P, Delberghe N, Le Bouar G, Miailhe AF, Hraiech S, Bironneau V, Sedillot N, Hoppe MA, Barbar SD, Calcaianu GD, Dellamonica J, Terzi N, Delpierre C, Gelinotte S, Rigaud JP, Labruyere M, Georges M, Binquet C, Quenot JP; RECOVIDS trial investigators. Influence of socioeconomic status on functional recovery after ARDS caused by SARS-CoV-2: a multicentre, observational study. BMJ Open. 2022 Apr 22;12(4):e057368. doi: 10.1136/bmjopen-2021-057368. PMID 35459672